CLINICAL TRIAL: NCT05390385
Title: Acceptability and Tolerability of Ketone Supplements and Their Effects on Capillary Beta-hydroxybutyrate Concentrations in Young Adults
Brief Title: Acceptability and Tolerability of Ketone Supplements and Effects of BHB Concentrations in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Eric P. Plaisance, Chairperson of the Department of Human Studies and Associate Professor of Exercise Physiology, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB-300009075
Record Dates: First submitted 2022-05-13; First posted 2022-05-25 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Exogenous Ketosis
Keywords: exogenous ketones; ketone supplementation; ketone monoester; ketone salt; tolerability; acceptability; beta-hydroxybutyrate

STUDY DESIGN:
Intervention Model Description: Participants will each undergo all five treatments, in randomized order. The five treatments include the control placebo, 5g of KE1, 10g of KE1, 5g of KE4, and 10g of KE4. There will be a minimum of two days washout period between treatments.
Who Masked: Participant, Investigator
Masking Description: Supplement packaging will be labeled with an alphanumeric code that is only understood by an individual who is not involved in the study. The participants and study team will both be blinded to the supplement being given.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control placebo (Placebo Comparator)
  Interventions: Other: Placebo drink
- KE1 5g (Experimental)
  Interventions: Dietary Supplement: KE1 5g
- KE1 10g (Experimental)
  Interventions: Dietary Supplement: KE1 10g
- KE4 5g (Experimental)
  Interventions: Dietary Supplement: KE4 5g
- KE4 10g (Experimental)
  Interventions: Dietary Supplement: KE 10g

INTERVENTIONS:
Dietary Supplement: KE1 5g — 5g of KE1 (KetoneAid, Falls Church, VA), diluted to 4 ounces
  Arms: KE1 5g
Dietary Supplement: KE1 10g — 10g of KE1 (KetoneAid, Falls Church, VA), equal to 4 ounces
  Arms: KE1 10g
Dietary Supplement: KE4 5g — 5g of KE4 (KetoneAid, Falls Church, VA), diluted to 4 ounces
  Arms: KE4 5g
Dietary Supplement: KE 10g — 10g of KE4 (KetoneAid, Falls Church, VA), diluted to 4 ounces
  Arms: KE4 10g
Other: Placebo drink — Flavor-matched control placebo drink (KetoneAid, Falls Church, VA), 4 ounces
  Arms: Control placebo

SUMMARY:
Assess the acceptability and tolerability of two different commercially available ketone supplements and determine their effects on capillary blood concentrations of the ketone beta-hydroxybutyrate and glucose in young adults.

DETAILED DESCRIPTION:
Past findings suggest that raising ketone concentrations through the use of a ketogenic diet (high-fat, moderate-protein, low-carbohydrate) is effective for preventing weight gain and decreasing appetite. However, strict adherence to this diet is difficult, and ending the diet can result in the regaining of body weight. Our group has investigated the effects of various ketone supplements in both rodents and humans. Past results of our group and that of our colleagues suggest that ketone supplements have the ability to increase ketone concentrations in the blood, decrease appetite, lower body weight, and maintain lean body mass. Exogenous ketones may serve as an alternative to the ketogenic diet by increasing concentrations of ketones without the need for adherence to a strict diet. However, little is known about ketone supplements as it relates to their tolerability and efficacy. For example, the taste of these supplements is unacceptable to some individuals and it is unclear if ketone supplements provide an adequate approach to raise and maintain circulating ketone concentrations as observed with the ketogenic diet. This information will be valuable before launching larger-scale human trials.

Ketone supplements (KE1 and KE4) will be obtained from KetoneAid (Falls Church, VA). Participants will be asked to drink (5g and 10g) of each supplement separated by at least 3 days. Capillary blood samples will be measured using a handheld device to measure circulating beta-hydroxybutyrate (BHB) and glucose concentrations while a questionnaire will be used to assess the acceptability and tolerability of the ketone supplements.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18-25 years of age
* In generally good health
* Able and willing to attend study visits (once every 3 days for ~2 weeks)
* BMI 18.5-29.9

Exclusion Criteria:

* Pregnant
* Has preexisting medical conditions, including Type 2 diabetes, heart disease, or cancer
* BMI ≥ 30

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Supplement tolerability and acceptability | 2 hours
  The ketone supplements being used have been described as having strong, disagreeable flavors. Therefore, the first outcome measure will be understanding how the flavors and gastrointestinal effects of both supplements may impact subjects. This outcome measure will be assessed by measuring the symptoms experienced, the time at which each symptom occurred, and the duration of each symptom using a scaled symptom questionnaire titled "Symptom Questionnaire." The questionnaire rates symptoms on an ordinal scale from absent, mild, moderate, to severe, with absent being the minimum value and better outcome, and severe being the maximum value and worst outcome. The questionnaire will assess the time that each symptom occurred, on a scale from immediately, one hour, and two hours after supplement consumption. The questionnaire will assess the duration of each symptom, on a scale of less than thirty minutes, one hour, and two hours after each symptom occurred.
Capillary beta-hydroxybutyrate concentrations | 2 hours
  Exogenous ketone supplements are now widely available at the commercial level, so it is important to understand the concentration-dependent effects of these supplements on circulating ketone concentrations, measured by concentrations of beta-hydroxybutyrate following a capillary blood fingerstick.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stubbs BJ, Cox PJ, Evans RD, Santer P, Miller JJ, Faull OK, Magor-Elliott S, Hiyama S, Stirling M, Clarke K. On the Metabolism of Exogenous Ketones in Humans. Front Physiol. 2017 Oct 30;8:848. doi: 10.3389/fphys.2017.00848. eCollection 2017. PMID 29163194